CLINICAL TRIAL: NCT01717521
Title: The Effects of Intravenous Administration of Ketamine on the Analgesia Nociception Index (ANI) Measured With the PhysioDoloris Device
Brief Title: Effects of IV Administration of Ketamine on the Analgesia Nociception Index (ANI) Measured With the PhysioDoloris
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Laurent Bollag, Assistant Professor, University of Washington
Other Study IDs: 42398
Record Dates: First submitted 2012-10-10; First posted 2012-10-30 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Monitoring, Intraoperative
Keywords: intraoperative monitoring; hysterectomy; robotic-assisted; abdominal gynecological surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study evaluates effects of the analgesic ketamine on ANI measurements (Anti Nociceptive Index)

DETAILED DESCRIPTION:
Researchers at the University of Washington are doing this study to find out if a commonly used anesthetic affects patients Analgesia Nociception Index (level of pain relief) during abdominal hysterectomy under general anesthesia.

The investigators will administer routine anesthesia care including Ketamine, a commonly used anesthetic, during the patients surgery. During the patients surgery, the investigators will monitor the patients level of pain relief using the PhysioDoloris monitor, which monitors the routinely used EKG monitor. Though not yet FDA approved, the PhysioDoloris is completely non-invasive and collects data from the EKG monitor.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II, or III
* 18 years or older
* Receiving GA with uncomplicated routine intubation
* Ability to provide informed consent
* English-speaking

Exclusion Criteria:

* Presence of coronary artery disease, cardiac arrhythmias, or ketamine allergy
* Patient refusal
* History of substance abuse
* Patients taking psychotropic and/or opiate drugs
* Having a history of psychiatric diseases or psychological problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing gynecological/abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bollag, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After institutional review board approval, this observational pilot study was conducted at the University of Washington Medical Center (UWMC). Twenty women, 18 years of age or older, of American Society of Anesthesiology Physical Status I-III scheduled for an abdominal hysterectomy under sevoflurane anesthesia were recruited.
Groups:
- Women, Scheduled for Abdominal Hysterectomy: Women 18 years of age or older, of American Society of Anesthesiology Physical Status I-III scheduled for an abdominal hysterectomy under general anesthesia
Period: Overall Study
Arm/Group | Women, Scheduled for Abdominal Hysterectomy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty women, 18 years of age or older, of American Society of Anesthesiology Physical Status I-III scheduled for an abdominal hysterectomy under sevoflurane anesthesia were recruited.
Groups:
- Women Scheduled for Abdominal Hysterectomies.: Inclusion criteria : >18yrs, ASA 1-3, Scheduled for abdominal hysterectomies under general anesthesia
Arm/Group | Women Scheduled for Abdominal Hysterectomies.
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Height [Mean (Standard Deviation); unit: cm] | 162.3 (9.6)
Weight [Mean (Standard Deviation); unit: kg] | 82.3 (35.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean ANI Changes After Intubation
Description: ANI stands for Analgesia Nociception Index. Its a dimension less number computed by a pain monitor ranging from 0-100. An index of 100 means absent pain, and the number decreases as pain increases. ANI was measured pre- and post- Intubation
Time Frame: Before vs after intubation
Population: This pilot study included 20 women undergoing abdominal hysterectomies
Measure: Mean (Standard Deviation); unit: index
Groups:
- Single Group: Participants undergoing abdominal hysterectomy under sevoflurane anesthesia
Arm/Group | Single Group
Number analyzed (Participants) | 20
index | 2.11 (20.11)

2. Primary Outcome: Mean ANI Changes 3 Min After Ketamine Bolus
Description: ANI was measured pre- and post- i.v. ketamine administration
Time Frame: Before vs 3 min after Ketamine adminstration
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Single Group
Number analyzed (Participants) | 20
index | 1.31 (15.26)

3. Primary Outcome: Mean ANI Changes 5 Min After Ketamine Bolus
Description: ANI was measured pre- and post- i.v. ketamine administration
Time Frame: Before vs 5 min after Ketamine adminstration
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Single Group
Number analyzed (Participants) | 20
index | 1.95 (17.67)

4. Primary Outcome: Mean ANI Changes After Skin Incision
Description: ANI was measured pre- and post- skin incision
Time Frame: Before vs after skin incision
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Single Group
Number analyzed (Participants) | 20
index | 13.65 (15.44)

5. Secondary Outcome: Mean BIS Changes After Intubation
Description: BIS was measured pre- and post-intubation.
  BIS, Bispectral index, is an indication of anesthesia depth and measured by a monitor during surgery (0-100 scale, range described below). Depth of sedation is calculated by measuring cerebral electric activity via an electroencephalogram (EEG).
  * 100-90: awake and responding appropriately to verbal stimulation
  * 80-70: responsive to loud commands or mild shaking
  * 60-40: unresponsive to verbal stimulus; general anesthesia obtained with a low chance for explicit recall
  * <40: deep hypnotic state; possible protective responses still intact
  * <20: burst suppression (EEG pattern characterized by cycles of high-voltage electrical movement alternating with cycles of no activity in the brain); respiratory drive is limited, but possible protective responses still intact
  * 0: totally suppressed EEG (flat line)
Time Frame: Before vs after intubation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 20
score on a scale | 7.25 (20.42)

6. Secondary Outcome: Mean BIS Changes 3 Min After Ketamine Bolus
Description: BIS was measured pre- and post-Ketamine administration.
  BIS, Bispectral index, is an indication of anesthesia depth and measured by a monitor during surgery (0-100 scale, range described below). Depth of sedation is calculated by measuring cerebral electric activity via an electroencephalogram (EEG).
  * 100-90: awake and responding appropriately to verbal stimulation
  * 80-70: responsive to loud commands or mild shaking
  * 60-40: unresponsive to verbal stimulus; general anesthesia obtained with a low chance for explicit recall
  * <40: deep hypnotic state; possible protective responses still intact
  * <20: burst suppression (EEG pattern characterized by cycles of high-voltage electrical movement alternating with cycles of no activity in the brain); respiratory drive is limited, but possible protective responses still intact
  * 0: totally suppressed EEG (flat line)
Time Frame: Before vs 3 min after Ketamine adminstration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 20
score on a scale | 3.3 (10.33)

7. Secondary Outcome: Mean BIS Changes After Skin Incision
Description: BIS was measured pre- and post-skin incision.
  BIS, Bispectral index, is an indication of anesthesia depth and measured by a monitor during surgery (0-100 scale, range described below). Depth of sedation is calculated by measuring cerebral electric activity via an electroencephalogram (EEG).
  * 100-90: awake and responding appropriately to verbal stimulation
  * 80-70: responsive to loud commands or mild shaking
  * 60-40: unresponsive to verbal stimulus; general anesthesia obtained with a low chance for explicit recall
  * <40: deep hypnotic state; possible protective responses still intact
  * <20: burst suppression (EEG pattern characterized by cycles of high-voltage electrical movement alternating with cycles of no activity in the brain); respiratory drive is limited, but possible protective responses still intact
  * 0: totally suppressed EEG (flat line)
Time Frame: Before vs after skin incision
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 20
score on a scale | 1.9 (5.71)

8. Secondary Outcome: Mean Heart Rate Change After Intubation
Description: Heart rate assessed by continuous pulse oximetry. Heart rate was measured pre- and post-intubation.
Time Frame: Before vs after intubation
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Single Group
Number analyzed (Participants) | 20
bpm | 5 (9)

9. Secondary Outcome: Mean Heart Rate Change 3 Min After Ketamine Bolus
Description: Heart rate was measured pre- and post- Ketamine administration
Time Frame: Before vs 3 min after Ketamine adminstration
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Single Group
Number analyzed (Participants) | 20
bpm | 2 (5)

10. Secondary Outcome: Mean Heart Rate Change After Skin Incision
Description: Heart rate was measured pre- and post-skin incision.
Time Frame: Before vs after skin incision
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Single Group
Number analyzed (Participants) | 20
bpm | 2 (6)

11. Secondary Outcome: Change in Mean Arterial Pressure After Intubation
Description: MAP or mean arterial pressure is the average blood pressure of an individual and is measured non-invasively during surgery. MAP was measured pre- and post-intubation.
Time Frame: Before vs after intubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 20
mmHg | 5.05 (19.99)

12. Secondary Outcome: Change in Mean Arterial Pressure After 3 Min After Ketamine Bolus
Description: MAP was measured pre- and post-ketamine administration
Time Frame: Before vs 3 min after Ketamine adminstration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 20
mmHg | 4.09 (18.52)

13. Secondary Outcome: Mean MAP Changes After Skin Incision
Description: MAP was measured pre- and post- skin incision.
Time Frame: Before vs after skin incision
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 20
mmHg | 13.5 (12.6)

14. Other Pre Specified Outcome: Average Ketamine Used
Description: Amount of Ketamine used during surgery
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Single Group
Number analyzed (Participants) | 20
mg | 41.3 (18)

ADVERSE EVENTS:
Groups:
- Single Group w Intervention: no adverse events were observed
Arm/Group | Single Group w Intervention
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes